CLINICAL TRIAL: NCT03306303
Title: Association Between Plasma Melatonin and No-reflow
Status: Completed | Type: Observational
Sponsor: Chinese PLA General Hospital (Other)
Responsible Party: Principal Investigator, Chen Wei Ren, MD, Doctor, Chinese PLA General Hospital
Other Study IDs: MelandNR
Record Dates: First submitted 2017-10-02; First posted 2017-10-11 (Actual); Last update posted 2017-10-11 (Actual); Status verified 2017-10

CONDITIONS: ST-segment Elevation Myocardial Infarction
Keywords: melatonin; STEMI; No-reflow
MeSH Terms: conditions — ST Elevation Myocardial Infarction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Biospecimen Retention: Samples Without DNA — melatonin, high-sensitivity C-reactive protein (hsCRP), superoxide dismutase levels
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Quartile 1 of plasma melatonin: Quartile 1 of plasma melatonin
- Quartile 2 of plasma melatonin: Quartile 2 of plasma melatonin
- Quartile 3 of plasma melatonin: Quartile 3 of plasma melatonin
- Quartile 4 of plasma melatonin: Quartile 4 of plasma melatonin

SUMMARY:
ST-segment elevation myocardial infarction (STEMI) is an acute manifestation of coronary heart disease, remaining a frequent cause of death. A better understanding of risk factors and pathogenic mechanisms underlying STEMI may help improve the prognosis and life quality of these patients. Melatonin is the chief indoleamine produced by the pineal gland, and a well-known antioxidant and free radical scavenger. Basic studies have showed that melatonin is associated with myocardial infarction and heart failure. However, no study has evaluated whether melatonin is associated with adverse clinical outcomes in STEMI patients.

ELIGIBILITY:
Inclusion Criteria:

a diagnosis of STEMI and needed PCI

Exclusion Criteria:

patients with cancer patients who used melatonin

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: PLA general hospital (PLAGH) is a large national tertiary-care center in the Beijing, China. The investigators enrolled all patients consecutively hospitalized in PLAGH, with a diagnosis of STEMI and needed PCI.
Sampling Method: Probability Sample
Enrollment: 1700 (Actual)
Dates: Start 2014-01-01 (Actual); Primary Completion 2017-10-01 (Actual); Study Completion 2017-10-01 (Actual)

PRIMARY OUTCOMES:
a change in the prevalence of no-reflow | mediately after percutaneous coronary intervention (PCI)
  Thrombolysis in myocardial infarction (TIMI) flow grade of <3 with a myocardial blush grade of 0-1 was defined as angiographic no-reflow

SECONDARY OUTCOMES:
in-hospital complications | up to 2 weeks after PCI
  defined as acute heart failure, atrial fibrillation, chest pain or recurrence of myocardial infarction, complete atrioventricular block, cerebrovascular disease, ventricular fibrillation or ventricular tachycardia
in-hospital major adverse cardiac or cerebrovascular events | up to 2 weeks after PCI
  the composite of death, nonfatal MI, or stroke

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Dominguez-Rodriguez A, Abreu-Gonzalez P, Arroyo-Ucar E, Reiter RJ. Decreased level of melatonin in serum predicts left ventricular remodelling after acute myocardial infarction. J Pineal Res. 2012 Oct;53(3):319-23. doi: 10.1111/j.1600-079X.2012.01001.x. Epub 2012 Apr 27. PMID 22537272
- [Background] Dominguez-Rodriguez A, Abreu-Gonzalez P, Reiter RJ. The potential usefulness of serum melatonin level to predict heart failure in patients with hypertensive cardiomyopathy. Int J Cardiol. 2014 Jun 15;174(2):415-7. doi: 10.1016/j.ijcard.2014.04.044. Epub 2014 Apr 15. No abstract available. PMID 24768380
- [Background] Tutuncu NB, Batur MK, Yildirir A, Tutuncu T, Deger A, Koray Z, Erbas B, Kabakci G, Aksoyek S, Erbas T. Melatonin levels decrease in type 2 diabetic patients with cardiac autonomic neuropathy. J Pineal Res. 2005 Aug;39(1):43-9. doi: 10.1111/j.1600-079X.2005.00213.x. PMID 15978056